CLINICAL TRIAL: NCT05586997
Title: Effect of Rapid Maxillary Expansion with Low Level Laser Therapy Versus Rapid Maxillary Expansion in Children with Posterior Cross Bite
Brief Title: Rapid Maxillary Expansion with Low Level Laser Therapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Collaborators: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Hend Salah ElSayed, Associate Professor, National Research Centre, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18055
Record Dates: First submitted 2022-10-16; First posted 2022-10-19 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-04

CONDITIONS: Crossbite; Malocclusion; Cross Bite; Maxillary Constriction
Keywords: bonded-Hyrax; Hyrax-expander; Maxillary constriction; Posterior cross bite; Rapid maxillary expansion
MeSH Terms: conditions — Malocclusion | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients will be masked by receiving sham LASER therapy in the control group. While, the outcome assessors will evaluate unidentified radiographic images and will have no knowledge of the intervention allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bonded Rapid Maxillary Expansion (Active Comparator): Bonded-hyrax with a 7mm expansion screw activated a full turn twice daily
  Interventions: Device: Bonded-Hyrax
- Bonded Rapid Maxillary Expansion and low-Level Laser (Experimental): Bonded-hyrax with a 7mm expansion screw activated a full turn twice daily with 10 sessions of Indium Gallium Arsenide Phosphoride (940nm) semiconductor diode laser
  Interventions: Device: Bonded-Hyrax; Combination Product: Bonded Rapid Maxillary Expansion and low-Level Laser therapy

INTERVENTIONS:
Device: Bonded-Hyrax — The expansion screw of the bonded-hyrax will be activated until the palatal cusps of the permanent maxillary first molars are opposing the buccal cusps of the permanent mandibular first molars
  Other Names: Rapid maxillary expansion (RME)
Combination Product: Bonded Rapid Maxillary Expansion and low-Level Laser therapy — Ten sessions of 0.5 watts for 20 seconds at 4 points along the mid-palatal suture
  Other Names: low level laser therapy (LLLT)
  Arms: Bonded Rapid Maxillary Expansion and low-Level Laser

SUMMARY:
The posterior crossbite is a common type of malocclusion that might affect the normal growth pattern. Early treatment is recommended by rapid maxillary expansion with different appliances. This line of treatment needs a sufficient retention period to decrease the rate of relapse. The low level laser therapy has been used to enhance tissue regeneration. This study aims to compare the effect of rapid maxillary expansion with low level laser versus rapid maxillary expansion in children with posterior cross bite malocclusions.

DETAILED DESCRIPTION:
This study aims to evaluate the effect of rapid maxillary expansion using the bonded Hyrax expander combined with low level Laser therapy versus rapid maxillary expansion alone. The investigators intend to recruit sixty subjects of both sexes, between the age of 7 and 14 years. Patients with posterior crossbites and patent Mid-palatal sutures will be randomized into one of the two groups of treatment. Full orthodontic records will be collected and the standard orthodontic radiographs will be replaced by cone beam computer tomographic images. The records will be taken before the maxillary expansion and after 6 months of retention. The skeletal, dentoalveolar, and soft tissue effects of the two interventions will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Posterior crossbite
2. Patent mid-palatal suture
3. Mixed dentition or early permanent teeth
4. Subjects who reported no medical conditions or prolonged medications

Exclusion Criteria:

1. Poor oral hygiene
2. Active periodontal disease
3. Craniofacial abnormalities
4. Previous orthodontic treatment
5. Any systemic disease or medication that might affect bone metabolism.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2019-05-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Inter-jugale width | six months of retention
  Horizontal distance between right and left Jugale points, in millimeters.
Buccal maxillary width | six months of retention
  Horizontal distance between the most lateral point on the right and left buccal alveolar plate at the level of the root trifurcation, in millimeters.
Bone density of the mid-palatal suture | six months of retention
  Average density of 200mm3 volume, in hounsfield units.

SECONDARY OUTCOMES:
Facial width | six months of retention
  Horizontal distance between right and left zygomatico-temporal points in millimeter.
Inter-infraorbitale width | six months of retention
  Horizontal distance between right and left infraorbitale points
Inter-lateral pterygoid width | six months of retention
  Horizontal distance between right and left lateral pterygoid points in millimeters
Nasal width | six months of retention
  Horizontal distance between right and left lateral nasale points in millimeters
Palatal maxillary width | six months of retention
  Horizontal distance between the most lateral point on the right and left palatal alveolar plate at the level of the root trifurcation, in millimeters.
Buccal alveolar bone thickness at the mesiobuccal root of the first maxillary permanent molar | six months of retention
  Horizontal distance between the most lateral point on the buccal alveolar plate opposite to the midpoint of the width of the mesiobuccal root of the upper permanent maxillary first molar at the level of the trifurcation
Buccal alveolar bone thickness at the distobuccal root of the first maxillary permanent molar | six months of retention
  Horizontal distance between the most lateral point on the buccal alveolar plate opposite to the midpoint of the width of the distobuccal root of the upper permanent maxillary first molar at the level of the trifurcation, in millimeter.
Palatal bone thickness | six months of retention
  Horizontal distance between the most lateral point on the right and left palatal alveolar plates at the level of the trifurcation of the upper permanent maxillary first molar.
Bi-gonial width | six months of retention
  Horizontal distance between right and left gonion points in millimeters
Inter-mental width | six months of retention
  Horizontal distance between right and left mental foramen in millimeters
alveolar tipping angle | six months of retention
  Angle between the tangent to palatal alveolar bone at right and left first molar and the mid sagittal plane
Dental tipping angle | six months of retention
  Angle between the line passing through palatal root apex and palatal cusp tip of the right and left first molar and the mid sagittal plane
Bone density of the nasal side of the Midpalatal suture | six months of retention
  Average density in hounsfield units.
Bone density of the oral side of the Midpalatal suture | six months of retention
  Average density in hounsfield units.
Upper airway dimension | six months of retention
  Volume of the upper airway in mm3
Intercanine width | six months of retention
  Distance between the right and left canine cusp tips.
Intermolar width | six months of retention
  Distance between the right and left central fossae of the permanent maxillary first molar
Inter-first premolar width | six months of retention
  Distance between the right and left first premolar buccal cusp tips.
Inter-second premolar width | six months of retention
  Distance between the right and left first premolar buccal cusp tips.
Pain score | Day 1 of appliance activation
  Visual Analogue Scale from 1-100. Zero denoting no pain and 100 denoting the worst pain imaginable
Day on which pain on activation stopped | Two weeks
  The day on which the patient reports no pain with appliance activation

CONTACTS AND LOCATIONS:
Overall Officials: Hend S ElSayed, PhD, Principal Investigator — National Research Centre, Egypt
Locations (1):
- Al-Azhar University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lagravere MO, Major PW, Flores-Mir C. Long-term dental arch changes after rapid maxillary expansion treatment: a systematic review. Angle Orthod. 2005 Mar;75(2):155-61. doi: 10.1043/0003-3219(2005)0752.0.CO;2. PMID 15825776
- [Background] Skondra FG, Koletsi D, Eliades T, Farmakis ETR. The Effect of Low-Level Laser Therapy on Bone Healing After Rapid Maxillary Expansion: A Systematic Review. Photomed Laser Surg. 2018 Feb;36(2):61-71. doi: 10.1089/pho.2017.4278. Epub 2017 Oct 25. PMID 29072861
- [Background] Kang Y, Rabie AB, Wong RW. A review of laser applications in orthodontics. Int J Orthod Milwaukee. 2014 Spring;25(1):47-56. PMID 24812743
- [Background] Baratieri C, Alves M Jr, de Souza MM, de Souza Araujo MT, Maia LC. Does rapid maxillary expansion have long-term effects on airway dimensions and breathing? Am J Orthod Dentofacial Orthop. 2011 Aug;140(2):146-56. doi: 10.1016/j.ajodo.2011.02.019. PMID 21803251
- [Background] Molen AD. Considerations in the use of cone-beam computed tomography for buccal bone measurements. Am J Orthod Dentofacial Orthop. 2010 Apr;137(4 Suppl):S130-5. doi: 10.1016/j.ajodo.2010.01.015. PMID 20381753